CLINICAL TRIAL: NCT06639178
Title: Phase II Trial to Determine the Effectiveness of an N-acetylcysteine and Urea-based Cream in Prevention of Capecitabine-induced HAND-foot Syndrome in Breast Cancer Patients
Brief Title: Effectiveness of an N-acetylcysteine and Urea-based Cream in Prevention of Capecitabine-induced HAND-foot Syndrome in Breast Cancer Patients
Acronym: HAND-TO-HAND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRO-2023-28
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DECLARAN cream (Experimental): Patients will apply of DECLARAN cream is the investigational product based on NAC and urea
  Interventions: Other: DECLARAN cream

INTERVENTIONS:
Other: DECLARAN cream — Patients will apply 1 mL of DECLARAN cream, as a single pressure dispensing (1 for hands, 1 for feet), 2 times/day on hands and feet, starting 3 days before the beginning of treatment with capecitabine and for the first 24 consecutive weeks of treatment.

SUMMARY:
Breast cancer (BC) is the most frequent tumour in women. To date, among the available treatments, the use of Capecitabine, an oral prodrug of fluorouracil, has been shown activity in different setting. In advanced disease, Capecitabine is often used as monotherapy in patients pretreated with anthracycline, taxane or both.

One of the most frequent toxicities reported by patients receiving capecitabine is hand-foot syndrome (HFS), with an incidence of grade 3 HFS of 28%. HFS, also known as palmar-plantar erythrodysesthesia syndrome, is initially characterized by palmoplantar numbness, tingling, or burning pain. These symptoms usually coincide with sharply demarcated erythema with or without edema, cracking, or desquamation. In advanced stages, blistering and ulceration may occur. Although HFS is not considered life threatening, it can be painful and interfere with daily activities, thusseriously compromising quality of life (QoL), therefore this toxicity is considered dose limiting.Moreover, consistent with the theory that Capecitabine and its metabolites induce an inflammatory effect, the use of COX-2 inhibitors is an emerging strategies, but more evidence are needed from largest study to confirm their efficacy.

Similarly, N-acetylcysteine (NAC), an antioxidant, mucolytic and nephroprotective agent, that affects pathways involved in inflammatory conditions and that has demonstrated to be effective in several dermatologic conditions, could be useful in the management of Capecitabine-induced HFS.

From this arises the present study that has the objective of evaluating the role of NAC plus urea-based cream in the prevention of Capecitabineinduced HFS in patient affected by breast cancer.

DETAILED DESCRIPTION:
Breast cancer (BC) is the most frequent tumour in women. To date, among the available treatments, the use of Capecitabine, an oral prodrug of fluorouracil, has been shown activity in different setting. In advanced disease, Capecitabine is often used as monotherapy in patients pretreated with anthracycline, taxane or both.

One of the most frequent toxicities reported by patients receiving capecitabine is hand-foot syndrome (HFS), with an incidence of grade 3 HFS of 28%. HFS, also known as palmar-plantar erythrodysesthesia syndrome, is initially characterized by palmoplantar numbness, tingling, or burning pain. These symptoms usually coincide with sharply demarcated erythema with or without edema, cracking, or desquamation. In advanced stages, blistering and ulceration may occur. Although HFS is not considered life threatening, it can be painful and interfere with daily activities, thusseriously compromising quality of life (QoL), therefore this toxicity is considered dose limiting.Moreover, consistent with the theory that Capecitabine and its metabolites induce an inflammatory effect, the use of COX-2 inhibitors is an emerging strategies, but more evidence are needed from largest study to confirm their efficacy.

Similarly, N-acetylcysteine (NAC), an antioxidant, mucolytic and nephroprotective agent, that affects pathways involved in inflammatory conditions and that has demonstrated to be effective in several dermatologic conditions, could be useful in the management of Capecitabine-induced HFS.

From this arises the present study that has the objective of evaluating the role of NAC plus urea-based cream in the prevention of Capecitabineinduced HFS in patient affected by breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women and men ≥18 years old
* Patients with diagnosis of breast cancer with stage I-III radically operated with residual disease post neoadjuvant treatment or stage IV
* Patients candidated for capecitabine in a post-neoadjuvant or metastatic setting treated with 2000-2500 mg/m2 d1-14 q21, or 1500 mg daily continuously (metronomic schedule)
* Patients who provided written informed consent

Exclusion Criteria:

* Patients previously treated with drugs that may have induced HFS
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol
* Pregnant, lactating, or breastfeeding, or intending to become pregnant during the study or within 60 days after the final dose of study treatmen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the role of NAC plus urea-based cream (DECLARAN) in the prevention of Capecitabine-induced HFS in patient affected by breast cancer. | up to 2 years
  Cumulative incidence of any grade HFS (according CTCAE vs 5.0,)

SECONDARY OUTCOMES:
To evaluate severe HFS | up to 2 years
  Cumulative incidence of grade 3 HFS according CTCAE vs 5.0
To evaluate the impact of HFS on patients' quality of life at 6 weeks | up to 2 years
  Cumulative incidence of summary values of patient reported outcome (PRO) assessed with HFS-14 at 6 weeks
To evaluate the impact of HFS on patients' quality of life at 12 weeks | up to 2 years
  Cumulative incidence of summary values of patient reported outcome (PRO) assessed with HFS-14 at 12 weeks
To evaluate the impact of HFS on patients' quality of life at 24 weeks | up to 2 years
  Cumulative incidence of summary values of patient reported outcome (PRO) assessed with HFS-14 at 24 weeks
To evaluate the safety of NAC plus urea-based cream | up to 2 years
  Frequecies of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Simon Spazzapan, MD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO) - IRCCS; Camilla Lisanti, MD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO) - IRCCS
Locations (2):
- Italy (2):
  - Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS, Aviano, Pordenone
  - Azienda Sanitaria Universitaria del Friuli Centrale (ASUFC), Udine